# ELECTRONIC CONSENT AND RESEARCH PARTICIPANT INFORMATION TITLE: "ImmuneRACE" – Immune Response Action to COVID-19 Events

**TITLE:** "ImmuneRACE" – Immune Response Action to COVID-19 Events

PROTOCOL NO.: ADAP-006

WIRB® Protocol #20200625

**SPONSOR:** Adaptive Biotechnologies Corporation

**INVESTIGATOR:** Jennifer Dines, MD

Adaptive Biotechnologies 1551 Eastlake Ave E

Suite 200

Seattle, Washington 98102

**United States** 

STUDY-RELATED

**PHONE NUMBER(S):** ImmuneRACE Toll Free Study Line (M-F 9 am – 8 pm EST)

(855)-419-3387

Study Doctor (206) 279-2486 Study Coordinator (206) 693-2032 Secure Fax Number (866) 623-4408

Secure Email

clinicalservices@adaptivebiotech.com

#### **SUMMARY**

You are being asked to be in a research study. This information sheet provides a detailed description of the study and how your participation would affect you.

- Being in a study is voluntary your choice.
- If you join this study, you may withdraw at any time.
- You may refuse to participate, or you may withdraw from the study at any time without penalty or loss of benefits to which you are otherwise entitled. This is not a treatment study. Options include not participating or participating in other research studies.
- You will not receive any direct benefits from being in this study, but you will be compensated for your participation.

AS MODIFIED Jul 28, 2020

# **PURPOSE OF THE STUDY**

Coronavirus disease is spreading rapidly throughout the world. The goal of the ImmuneRACE study is to learn about a patient's immune response to the virus. Your blood will be collected for this study. Data from blood samples will be analyzed to better understand the immune system. De-identified data will be shared with the research community with the potential goal of understanding the immune system response to coronavirus disease to aid in helping develop better tests and treatment for coronavirus disease, and the potential of developing a diagnostic test from data collected in this study. The tests used are investigational. You will not receive the results of any tests.

The ImmuneRACE study is part of Adaptive's T-cell receptor (TCR)-Antigen Map project, a partnership with Microsoft to use artificial intelligence (AI) and machine learning to accelerate our ability to map how the immune system responds to diseases.

#### **SCOPE OF YOUR PARTICIPATION**

Your participation will consist of completing a questionnaire, a blood draw, and a nose or throat swab. Standard blood draws will be performed by inserting a needle into a vein in your arm (venipuncture). Blood will be collected in volumes of approximately 1-4 tablespoons. The nose or throat swab will be collected by rubbing the swab on the inside of your nose or throat.

Demographic information, information relating to coronavirus disease, and medical information, such as, but not limited to, medications and other health conditions, that may impact study results will be collected from you by a study questionnaire and review of your relevant medical records. In some cases, we may require you to provide a wet ink signature on a Health Insurance Portability and Accountability Act (HIPAA) form to be shared with the provider network. We will ask you to provide diagnostic test results performed for coronavirus disease if performed and available. These test results include results from your nose or throat swab (PCR) testing and antibody test results. Diagnostic test results can be provided to the secure email or secure fax number listed above.

By consenting to be in the ImmuneRACE study you agree that you are willing to provide your blood, undergo a nose or throat swab for this research, complete a questionnaire, provide diagnostic test results for coronavirus disease if performed, and allow access to your health information. You will be eligible for receipt of a \$50 gift card upon completion of your participation in the study. Completion is defined as receipt of blood sample, nose or throat swab and completed questionnaire (all questions answered).

The data collected from this study from your blood cells, nose or throat swab, and health information will be stored with a code, not with your name. Any link between the code and your name will be kept separately and will only be available to the study doctor and key members of the study team.

IRB APPROVED AS MODIFIED Jul 28, 2020

Your samples collected in the ImmuneRACE study will be used and stored until the sample is exhausted (there is no sample remaining). It is possible that your blood and nose or throat swab sample may be used to run additional tests that diagnose or support the diagnosis of coronavirus disease in addition to other diseases. Future research using your sample may lead to the development of commercial products. You will not share in any profits that the research may produce.

Physical risks associated with drawing blood, include: soreness at the site of puncture, bruising, and in rare case, infection of the blood draw site, fainting, nerve or tendon damage. Physical risks associated with a nose or throat swab include: a very small risk of bleeding when swabbing the inside of your nose or throat (mucosal membranes). Participation in research also involves a risk of loss of confidentiality. All studies may involve unforeseeable risks.

In addition to your participation in the ImmuneRACE study, you have the option to consent to participating in up to four additional blood draws and up to 4 web-based questionnaires about your symptoms and medical information relating to coronavirus disease over a two-month time period. You can revoke your consent at any time. You can complete the ImmuneRACE study without consenting to or completing additional blood draws and questionnaires. Each additional blood draw will be in volumes of approximately 1-4 tablespoons. You will be given an additional \$50 gift card after completing each additional blood draw and questionnaire concerning your symptoms and medical information about coronavirus disease.

#### OTHER IMPORTANT INFORMATION

- Dr. Jennifer Dines is an employee of the Sponsor and does possess stock options from this company. Please feel free to ask any further questions you might have about this matter.
- You will be told about any new information that might change your decision to be in this study. You may be asked to sign a new consent form if this occurs.
- You may be removed from the research by the study doctor or sponsor if it is in your best interest, you do not consent to continue in the study after being told of changes in the research that may affect you, or for any other reason.
- We will not return individual results from this study, nor give the results to your doctor or put them in your medical record.
- Neither you nor your insurance company will be billed for your participation in this study.

For additional details on "What to Expect with Participation in a Research Study", please refer to FAQ [hyperlink to FAQ].

#### **AUTHORIZATION TO USE AND DISCLOSE INFORMATION FOR RESEARCH PURPOSES**

An important part of this Consent is your authorization for the study doctor and study team to use and disclose the personal information about you that will be collected for purposes of the study (referred to as "information" below).

#### Who else might get this information besides the study doctor and study team?

The sponsor of this research ("Sponsor"), meaning Adaptive Biotechnologies and any persons or companies that are:

- working for or with Adaptive Biotechnologies such as study partners (Microsoft, LabCorp/Covance and Illumina),
- or any affiliates owned by Adaptive Biotechnologies.

Study information may also be reviewed and/or copied for research or regulatory purposes by Western Institutional Review Board® (WIRB®).

### Why will this information be used and/or given to others?

- To do the research, to study the results, and to see if the research was done right.
- To permit study team members, (for example, the local phlebotomist (person drawing blood and collecting nasal or throat swab)) to contact you directly to schedule an appointment, ask questions relating to your symptoms and diagnosis of coronavirus during the visit, and grant access to your electronic medical records as necessary.
- These individuals will have access to your name, sex, address, phone number and study number. Your information will be maintained in a secure system.

# May I withdraw or revoke (cancel) my authorization for use and disclosure of my health information?

Yes, you may withdraw (revoke) your permission to use and disclose your health information at any time. You do this by sending written notice to the study doctor at the address shown on page 1. However, if you withdraw your permission for use and disclosure of your health information, you will not be able to stay in this study. Also, although withdrawing your permission will prevent further uses and disclosures of your health information, it will not invalidate uses and disclosures that have already been made at the time the permission is withdrawn. This permission will be good until December 31, 2060.

#### Is my health information protected after it has been given to others?

Every effort will be made to ensure confidentiality of Protected Health Information (PHI) in accordance with HIPAA. There is a risk that your information will be given to others without your permission, but disclosures of your health information will be very limited, as described above. If the results of this research study are presented at meetings or in publications, your identity will not be included in the information that is disclosed. Government agencies such as

IRB APPROVED AS MODIFIED Jul 28, 2020

the FDA or staff sometimes review studies such as this one to make sure they are being done safely and legally. If a review of this study takes places, your records may be examined. The reviewers will protect your privacy. The study records will not be used to put you at legal risk.

#### **QUESTIONS**

If you have questions, concerns, or complaints, or think this research has hurt you or made you sick, talk to the research team at the phone number listed above on the first page.

This research is being overseen by an Institutional Review Board ("IRB"). An IRB is a group of people who perform independent review of research studies. You may talk to them at (800) 562-4789, help@wirb.com if:

- You have questions, concerns, or complaints that are not being answered by the research team.
- You are not getting answers from the research team.
- You cannot reach the research team.
- You want to talk to someone else about the research.
- You have questions about your rights as a research subject.

# **ELECTRONIC CONSENT**

I have read this information sheet thoroughly. I freely consent to be in this research study.

I authorize the use and disclosure of my health information (collected as part of this research) to the parties listed in the authorization section of this consent for the purposes described above.

By clicking "ACCEPT", I agree to participate in the ImmuneRACE study.

In addition, I have made the optional choice marked below. I know that I can take still take part in the ImmuneRACE Study, even if I answer 'no' to the following option(s).

1. I elect to have up to four additional blood draws and complete up to four additional questionnaires relating to my symptoms and medical care relating to coronavirus disease as part of this study. I know that I can revoke (cancel) my approval for this at any time. In addition, I know that I can still complete the ImmuneRACE study without doing additional blood draws or questionnaires.

Select "YES" or "NO"

2. Researchers at Adaptive Biotechnologies may contact me about offers to take part in future Adaptive Biotechnologies' research. There will be a new consent process for that study. I can decide then to take part or not take part.

Select "YES" or "NO"

3. Employees at Adaptive Biotechnologies may contact me about other opportunities outside of a research study, such as sharing my story with my permission. I understand that Adaptive Biotechnologies may publish this content online and in print materials, and it may be revised and used in part or in its entirety.

Select "YES" or "NO"